CLINICAL TRIAL: NCT00408460
Title: A Phase II Study of Intermittent Gleevec® (Imatinib Mesylate) and Weekly Paclitaxel in Patients Aged 70 or Older With Advanced Non-Small Cell Lung Cancer
Brief Title: Imatinib Mesylate and Paclitaxel in Treating Older Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Renato Martins, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6137; NCI-2010-00420 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-01

CONDITIONS: Malignant Pleural Effusion; Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Imatinib Mesylate; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (enzyme inhibitor, chemotherapy) (Experimental): Patients receive paclitaxel IV on days 3, 10, and 17 and imatinib mesylate PO QD on days 1-4, 8-11, and 15-18. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Drug: paclitaxel

INTERVENTIONS:
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol

SUMMARY:
This phase II trial is studying how well giving imatinib mesylate together with paclitaxel works in treating older patients with stage IIIB or stage IV non-small cell lung cancer. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving imatinib mesylate together with paclitaxel may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the clinical efficacy of the combination of weekly paclitaxel and intermittent imatinib in elderly patients with advanced non-small cell lung cancer.

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of the combination of weekly paclitaxel and intermittent imatinib in elderly patients with advanced non-small cell lung cancer.

II. To collect paraffin tissue blocks for a companion project evaluating the expression of platelet derived growth factor (PDGF) by original tumor specimens, and its relationship to response rate and survival.

OUTLINE:

Patients receive paclitaxel intravenously (IV) on days 3, 10, and 17 and imatinib mesylate orally (PO) once daily (QD) on days 1-4, 8-11, and 15-18. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of non-small cell lung cancer
* At least one site of measurable disease, as defined by the modified RECIST criteria
* Stage IIIB with pleural effusion or Stage IV disease; includes patients who received surgery alone for early stage disease, now in relapse with advanced disease; staging is according to the American Joint Committee on Cancer classification scheme, 6th edition
* Total bilirubin < 1.25 x upper limit of normal (ULN)
* Baseline absolute neutrophil count >= 1500/uL
* Baseline platelet count >= 100,000/uL
* ECOG Performance Status 0, 1 or 2 at the time of informed consent
* Written, voluntary consent
* Patients with reproductive potential must use an acceptable contraceptive method, such methods include: 1) Male hormonal contraception; 2) Partner without reproductive potential, including post-menopausal status or history of tubal ligation; 3) Partner with intrauterine device (IUD) or contraceptive vaginal ring; 4) Partner takes oral contraceptive pill, wears contraceptive patch, or has contraceptive implant; 5) Routine use of barrier method, such as condoms or diaphragm, during sexual intercourse
* AST and ALT =< 2.5 x ULN
* Creatinine =< 1.5 x ULN

Exclusion Criteria:

* Uncontrolled brain metastasis; patients with known brain metastasis must have completed treatment with surgery, radiation or both; in addition, they must be off corticosteroids
* Symptomatic neuropathy (Grade 2 or higher)
* Prior chemotherapy for advanced non-small cell lung cancer (Prior adjuvant, neoadjuvant, or chemoradiotherapy for NSCLC is permitted, provided at least 6 months elapsed prior to documented metastatic recurrence)
* Patient is < 5 years free of another primary malignancy, except: a) if the other malignancy is basal cell carcinoma or cervical carcinoma in situ or b) if the other primary malignancy is not considered clinically significant and is requiring no active intervention
* Prior radiation therapy to > 25% of bone marrow
* Grade III/IV congestive heart failure, as defined by NYHA criteria, or myocardial infarction within 6 months
* Any serious or uncontrolled concomitant disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study
* Patient has known chronic liver disease, e.g., diagnosis of chronic active hepatitis or cirrhosis
* Major surgery two weeks prior to study treatment
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent
* Any condition requiring continuous administration of systemic corticosteroids
* The patient is on therapeutic anti-coagulation with warfarin
* The administration of any other anticancer agents including chemotherapy and biologic agents is NOT permitted
* The use of other concurrent investigational drugs is not allowed
* Participants in this study must avoid grapefruit juice or other grapefruit-containing products for the duration of treatment with imatinib

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-02; Primary Completion 2010-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato Martins, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients that were aged 70 years and above that had never received treatment for metastatic NSCLC were approached for study participation.
Groups:
- Treatment (Enzyme Inhibitor, Chemotherapy): Patients receive paclitaxel IV on days 3, 10, and 17 and imatinib mesylate PO QD on days 1-4, 8-11, and 15-18. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  imatinib mesylate: Given PO
  paclitaxel: Given IV
  immunohistochemistry staining method: Optional correlative studies
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor, Chemotherapy)
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor, Chemotherapy)
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 34
Age, Continuous [Median (Full Range); unit: years] | 75 [70 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete and Partial Responses) as Assessed by RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Baseline, Week 4 of courses 2, 4 and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Enzyme Inhibitor, Chemotherapy)
Number analyzed (Participants) | 34
Participants | 11

2. Secondary Outcome: Time to Tumor Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Baseline and every 2 months post treatment until the date of first documented tumor progression or date of death from any cause, whichever came first, assessed up to 5 years.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Enzyme Inhibitor, Chemotherapy)
Number analyzed (Participants) | 34
months | 3.6 [0.5 to 103]

3. Secondary Outcome: Overall Survival
Time Frame: Every 3 months for 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Enzyme Inhibitor, Chemotherapy)
Number analyzed (Participants) | 34
months | 7.3 [0.5 to 60]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of imatinib mesylate through to the last dose of imatinib mesylate, an average of 6 months.
Description: Only grade 3 and higher adverse events were collected with the following exceptions. Any grade neuropathy or edema and any other adverse event that required a dose reduction or dose delay.
Arm/Group | Treatment (Enzyme Inhibitor, Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 14/34
Other Adverse Events (participants affected / at risk) | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor, Chemotherapy) (N=34)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
cardiac arrest (Cardiac disorders) | 3 (3)
CHF exacerbation (Cardiac disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder Stone (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor, Chemotherapy) (N=34)
anemia (Blood and lymphatic system disorders) | 3 (3)
leukopenia (Blood and lymphatic system disorders) | 4 (4)
neutropenia (Blood and lymphatic system disorders) | 7 (7)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Edema (General disorders) | 8 (8)
acute kidney injury (Renal and urinary disorders) | 4 (4)
hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Foot Drop (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 10 (10)
Syncope (Nervous system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
increased pain (Nervous system disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Kidney stone (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes